CLINICAL TRIAL: NCT01848587
Title: Trial of Acupuncture Pelvic and Low Back Pain in Pregnancy (TAPPP)
Brief Title: Trial of Acupuncture Pelvic and Low Back Pain in Pregnancy (Medical and Economical Assessment)
Acronym: GAME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P111001
Record Dates: First submitted 2013-03-06; First posted 2013-05-07 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2014-06

CONDITIONS: Disorder of Pregnancy
Keywords: Pregnancy; Acupuncture; Pelvic and low back pain; Impairment; Economic evaluation
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture (Experimental): 5 acupuncture sessions over a 4 week period plus standard treatment
  Interventions: Other: acupuncture
- usual care (Active Comparator): standard treatment (pregnancy belt, behavioral recommendations, exercises, pain killers as prescribed by usual health care professional)
  Interventions: Other: usual care

INTERVENTIONS:
Other: acupuncture
  Arms: acupuncture
Other: usual care
  Arms: usual care

SUMMARY:
Pelvic girdle and low back pain are common in pregnancy, and cause severe impairment in 10% of women. Our hypothesis is that offering acupuncture in addition to standard care would reduce pain and impairment throughout pregnancy. 300 pregnant women from 5 maternity units will be randomized over a 3 year period to receive standard care or standard care plus acupuncture. Main outcome will be the number of days during pregnancy with maximum pain ≤ 4/10. Secondary outcomes will compare groups for an impairment score and for direct and indirect costs.

DETAILED DESCRIPTION:
Background. Pelvic and low back pain (PLBP) affects 30% of pregnant women for weeks or months, causing severe impairment in 10% of women. Standard treatment, based on pain killers, postural recommendations, exercises, is of limited value. Previous trials showed that adding acupuncture to standard treatment reduces pain and impairment in the short run.

Hypothesis Providing acupuncture to pregnant women with PLBP could reduce pain and impairment throughout pregnancy, thus reducing other direct and indirect cots related to PLBP.

Primary Outcome. Number and % of days during pregnancy with maximum pain ≤ 4/10.

Secondary Outcomes. Pain scale 4 weeks after inclusion, mean Oswestry disability score between inclusion and delivery, direct costs related to pregnancy care and pain management, indirect costs related to impairment throughout pregnancy and the immediate postpartum.

Method. Multicenter randomized trial with parallel groups. Intervention: 5 acupuncture sessions over 4 weeks, plus standard treatment. Controls: standard treatment.

Analysis per pregnancy Follow up: logbook kept by he patient plus analysis of obstetrical records. Number of patients: 300 Inclusion criteria: singleton uncomplicated 16-34 weeks pregnancy, with PLBP > 4/10 Exclusion criteria Obstetrical complication other than PLBP, contra indication to acupuncture, sciatica, maternal age < 18, no health insurance.

Duration. Overall duration: 3 years and 6 months, inclusions over 3 years. Duration of inclusion per patient: 2-26 weeks Number of participating centers 5

ELIGIBILITY:
Inclusion Criteria:

* singleton uncomplicated 16-34 weeks pregnancy, with PLBP > 4/10

Exclusion Criteria:

* Obstetrical complication other than PLBP,
* contra indication to acupuncture,
* sciatica
* maternal age < 18
* no health insurance.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number and % of days during pregnancy with maximum pain ≤ 4/10. | at 4 weeks
  daily recording on logbook (self assessment)

SECONDARY OUTCOMES:
Mean Oswestry disability score | during pregnancy
Number and % of days with maximum pain ≤ 4/10. | during pregnancy
direct and indirect costs | during pregnancy
  direct costs related to pregnancy care and pain management, indirect costs related to impairment throughout pregnancy and the immediate postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dommergues, Md, PhD, Principal Investigator — APHP
Locations (1):
- Centre d'Investigation Clinique Paris Est - Hôpital Pitié Salpêtrière, Paris, France

REFERENCES:
- [Result] Nicolian S, Butel T, Gambotti L, Durand M, Filipovic-Pierucci A, Mallet A, Kone M, Durand-Zaleski I, Dommergues M. Cost-effectiveness of acupuncture versus standard care for pelvic and low back pain in pregnancy: A randomized controlled trial. PLoS One. 2019 Apr 22;14(4):e0214195. doi: 10.1371/journal.pone.0214195. eCollection 2019. PMID 31009470